CLINICAL TRIAL: NCT01743326
Title: Percutaneous Radiofrequency Denervation of the Cervical Facet Joints Compared With Cervical Medial Branch Block of the Facet Joints for Patients With Chronic Degenerative Neck Pain : A Prospective Randomized Clinical Study
Brief Title: RFD Versus Cervical Medial Branch Blocks in Chronic Degenerative Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: METC 12-2-031
Record Dates: First submitted 2012-11-21; First posted 2012-12-06 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Facet Joint Arthritis; Pain; Radiofrequency Denervation
Keywords: Zygapophyseal Joint
MeSH Terms: conditions — Pain | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFD-group (Experimental): Radio Frequency Denervation
  Interventions: Procedure: Radio Frequency Denervation; Procedure: Local Anesthesia
- Local Anesthesia-group (Active Comparator): Local Anesthesia-group
  Interventions: Procedure: Local Anesthesia

INTERVENTIONS:
Procedure: Radio Frequency Denervation
  Arms: RFD-group
Procedure: Local Anesthesia

SUMMARY:
Rationale: the facet joints are an important pain generator in chronic neck pain. The beneficial effect of radio frequency treatment (RFD) of the cervical facet joints has been described in a Randomized Clinical Trial (RCT) in patients with Whiplash Associated Disorders. In patients with degenerative neck complaints a positive effect has been described in observational studies. Given this positive effect performing a RCT of RFD in this patient population is indicated.

Objective: to evaluate the effect of Radio Frequency treatment in patients with chronic degenerative neck pain.

Study design: prospective, randomized, double blinded clinical trial. Study population: patients older than 25 years, referred to the University Pain Center of Maastricht and the Pain Center of Amphia hospital Breda, with chronic axial neck pain.

Intervention: patients with at least 3 months of neck pain without radiation to the arm (only radiation beyond the shoulder) will be randomized in 2 groups. The first group (RFD + local anesthesia-group=intervention group) will receive RF treatment adjacent to the medial branch innervating the cervical facet joints after the application of bupivacaine 0.5 ml (0.25%). The second group (local anesthesia-group=control group) will only receive the application of 0.5 ml bupivacaine (0.25%) adjacent to the medial branch. The only difference between the two groups is the RF-denervation of the medial branches.

Main study parameters/endpoints: the primary research question is to evaluate the extent of pain reduction induced by RF treatment (RFD + local anesthesia-group=intervention group) compared with the local anesthesia-group(control group.

Following evaluation tools are used : Numeric Rating Scale (NRS), Patient global Impression of Change on a 7 point Likert Scale (PGIC), consumption of pain medication (MQS), Patient Specific Functional Scale, Quality of life scale (RAND 36), Hospital Anxiety and Depression scale (HADS), and Neck Disability Index (NDI, Dutch version).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients in the RFD + Local Anesthesia-group and Local Anesthesia-group will undergo a physical examination before and 6 weeks after the intervention, by an independent third party, this will be repeated at 3 and 6 months if abnormalities are observed. At each of these time points the patients will receive questionnaires to fill out. A puncture of a blood vessel is possible, diagnosed by injection of contrast, for which repositioning of the needle is needed. Should accidental intravascular injection of local anesthetic occur, the dose used is low and reports show that intravascular injection of bupivacaine 2,5 mg does not pose clinical problems. The dura can be punctured; as a consequence contrast will flow in the cerebrospinal fluid. The procedure will be stopped and repeated after a few days. In theory a lesion of the nerve root is possible, but the needles are designed to avoid this, this complication has not been seen since more than 10 years. Up till now, a transient pain is occasionally described after the RF treatment. No hypesthesia or motor complications were reported. Since the risks of RF treatment are reported low and more related to needle placement there is no difference in risk and burden between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age > 25 year
* Signs of degeneration on lateral X-ray
* Cervical facets to be treated between C2 and C7
* Pain for at least 3 months and conservative treatment medication (=paracetamol, Non-Steroidal anti-inflammatory Drugs (NSAID) and/or physical therapy) prior to referral to the pain clinic
* Neck pain on a Numeric Rating Scale ≥ 5

Exclusion Criteria:

* Radiation beyond the shoulder/radicular pain
* Shoulder pain/pathology
* The complaints are directly related to traumatic event e.g. Whiplash (WAD)
* Patient is pregnant, or pregnancy is suspected
* Patient has a cardiac pacemaker, automatic defibrillator or any leads in the neck area
* Allergy to contrast media or drugs to be used in the procedure
* History of anterior fusion at the cervical level to be treated
* Patient is simultaneously participating in another device or drug study related to cervical pain.
* Patient has a spinal fracture, tumor or infection.
* Patient has a central cord lesion in the cervical spine
* Neurologic deficit
* Evidence of disc herniation (extruded, sequestered on MRI imaging)

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Mean pain intensity measured on a 11-point Numeric Rating Scale (NRS). | Baseline, 6 months
Patient Global Impression of Change according to a 7-point Likert scale (PGIC). | Baseline, 6 months
Changes in use of pain medication according to the Medication Quantification Scale (MQS). | Baseline, 6 months
Changes in the Neck Disability Index scale (NDI). | Baseline, 6 months

SECONDARY OUTCOMES:
Changes in quality of life and differences between groups by means of RAND 36. | Baseline, 6 months
Improvement in functionality measured by the Patient Specific Functional Scale. | Baseline, 6 months
Change in physical/neurological examination parameters. | Baseline, 6 months
Change in employment status. | Baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van Kleef, Prf. MD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands